CLINICAL TRIAL: NCT03587233
Title: Physical Activity Level and Gender-differences of Adults in Different Professional Status
Brief Title: Are Women With Higher Professional Status More Sedentary Compared to Men?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Habibe Serap Inal, Prof.Dr., Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Bahcesehir
Record Dates: First submitted 2018-06-26; First posted 2018-07-16 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Professional Role; Physical Activity; Obesity; Education; Body Composition
Keywords: Weight status; Body mass index; Physical activity level; Lifestyle behaviour
MeSH Terms: conditions — Motor Activity; Obesity | interventions — Restraint, Physical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Women with higher professional status (Active Comparator): Women with higher professional status working in the Universities as academicians will be assessed regarding to their physical condition as weight status, BMI, waist and neck circumference, body composition and physical activity level, hand and pinch grip power to perform the intervention of physical assessment.
  The Turkish version of the 'International Physical Activity Questionnaire (IPAQ)-Short Form', the analyses of body composition will used to perform the intervention on the physical activity level. The outcomes of women with higher professional status will be compared with the other arms/groups as before and after the training program on exercise and healthy eating habits.
  Interventions: Behavioral: Physical assessment; Device: Analyses of body composition; Behavioral: physical activity level assessment
- Women with lower professional status (Active Comparator): Women with lower professional status in the cleaning companies will be assessed regarding to their physical condition as weight status, BMI, waist and neck circumference, body composition and physical activity level, hand and pinch grip power to perform the intervention of physical assessment.
  The Turkish version of the 'International Physical Activity Questionnaire (IPAQ)-Short Form', the analyses of body composition will used to perform the intervention on the physical activity level. The outcomes of women with lower professional status will be compared with the other arms/groups as before and after the training program on exercise and healthy eating habits.
  Interventions: Behavioral: Physical assessment; Device: Analyses of body composition; Behavioral: physical activity level assessment
- Men with higher professional status (Active Comparator): Men with higher professional status working in the Universities as academicians will be assessed regarding to their physical condition as weight status, BMI, waist and neck circumference, body composition and physical activity level, hand and pinch grip power to perform the intervention of physical assessment.
  The Turkish version of the 'International Physical Activity Questionnaire (IPAQ)-Short Form', the analyses of body composition will used to perform the intervention on the physical activity level. The outcomes of men with higher professional status will be compared with the other arms/groups as before and after the training program on exercise and healthy eating habits.
  Interventions: Behavioral: Physical assessment; Device: Analyses of body composition; Behavioral: physical activity level assessment
- Men with lower professional status (Active Comparator): Men with lower professional status working in the cleaning companies will be assessed regarding to their physical condition as weight status, BMI, waist and neck circumference, body composition and physical activity level, hand and pinch grip power to perform the intervention of physical assessment.
  The Turkish version of the 'International Physical Activity Questionnaire (IPAQ)-Short Form' and the analyses of body composition will used to perform the intervention on the physical activity level. The outcomes of men with lower professional status will be compared with the other arms/groups as before and after the training program on exercise and healthy eating habits.
  Interventions: Behavioral: Physical assessment; Device: Analyses of body composition; Behavioral: physical activity level assessment

INTERVENTIONS:
Behavioral: Physical assessment — Besides the demographic features of the participants, the interventions on physical assessment will be performed including weight in kilogram and height in meter; and weight and height will be combined to report body mass index in kg/m2. The waist circumference will be measured to understand the central fattening from costal margins or above umbilicus in cm. If it is measured above 95cm for men and 80cm for women is considered as higher than normal; if higher than 110cm for men and 88cm for women is considered as having risks for obesity, diabetes, cardiovascular diseases etc. Hand and pinch grip power will be assessed. It the elbow is in extension upper extremity power, and if it is flexed at 90 degree and forearm is supported on the table handgrip power is to assess.
Device: Analyses of body composition — The analyzes of body composition will be measured with bioelectrical impedance analysis method by a body composition analyzer.
Behavioral: physical activity level assessment — The physical activity level will be assessed through the intervention titled with the Turkish version of the 'International Physical Activity Questionnaire-Short Form'. It consists of seven questions searching for the amount of walking and low, moderate and high intensity physical activities as total time in minutes per day and frequency in days per week. Sitting, as a sedentary behavior, will be evaluated separately. The scores will be achieved by the multiplication of the minutes, days and metabolic equivalent time values in a week, and over the last 7 days. Walking score and total weekly walking duration will be calculated as medium and vigorous; the physical activity level will be classified as low, moderate and high level activity.

SUMMARY:
It is aimed to understand the gender differences on factors affecting the resting metabolic rate of people in different professional status.

The relation between daily and weekly walking and sitting time, body mass index (kg/m2), Ponderal Index (kg/cm), waist-to-hip ratio of the participants will be searched. In this context, the demographic data (age, gender, neck and waist circumference (cm), occupation, education level) of the participants will be gathered with a questionnaire, specifically prepared for this study. The body composition analyses and International Physical Activity Level Questionnaire (IPAQ), Healthy Eating Index (HEI) will also be used to understand their body composition, physical activity level and eating habits, respectively. The data will be compared to understand the effects of education level and type of occupation on their physical activity level, as well as, the effects of trainings on adapting healthy behaviour of the participants as physical activity, healthy eating habits in relation to gender and professional status.

DETAILED DESCRIPTION:
Being overweight and obese are becoming serious health care problems in developed countries as well as in Turkey. Both are associated with severe health problems as increased risk of heart disease, hypertension, diabetes, dyslipidemia, stroke, gallbladder disease, osteoarthritis, sleep apnea, respiratory and renal problems, and certain types of cancer. The behavioral and environmental factors (i.e. sedentary lifestyles combined with excess energy intake, unhealthy diet, low level of education and poverty) are primarily responsible for the dramatic increase of obesity. In Turkey, the prevalence of obesity has increased by 65% among men and 30% among women during the 90's. According to the recent findings of The National Household Research the incidence of being overweight was 31.35% and obese was 12.2% among those above 18 years. This was 28.93% and 14.59% in females and 33.64% and 9.70% in males, respectively. It was also reported that the incidence of being overweight had a tendency to increase linearly by age: 2.53% between 18-24 years, 7.96% between 25 - 34 years, 15.57% between 35-44 years, 22.61% between 45-54 years, 22.55% between years 55 - 64 years. This increase in obesity with aging may not be only due to the decrease in the fat-free mass but also due to an impaired ability to regulate the energy balance with age. Therefore, the age-related decline in basal metabolic rate, which is also related to the reduction in fat-free mass may alter the energy balance and contribute to weight gain. Thus, physical activity is essential for obese subjects in order to maintain or to increase their basal metabolic rate as well as their daily energy expenditure to enhance their weight loss.

Therefore, regular physical exercise may be considered as an effective tool to increase the resting metabolic rate by improving the muscle mass. However, the modern life, equipped with technological support, has eventually decreased the amount of daily physical activities in household tasks, transportation or in work environments. As Kirk and Rhodes stated the positions of higher professional status are more likely to engage in sedentary work-related behavior (i.e. sitting) compared to those working in positions of lower professional status (i.e. manual labor). Additionally, male were more likely to be employed in blue-collar or high-manual-labor positions that require high physical activity compared to women. The women mostly prefer non-occupational and non-leisure activities; for instance house-work. It is also reported that low level physical activity habit is higher among people having office work and living in the cities in Turkey.

Therefore, we have aimed to evaluate the physical activity level, physical status and the eating habits of the people in higher or lower professional statuses, and observe the gender differences.

ELIGIBILITY:
Inclusion Criteria:

* High status Professionals in both gender(white collars)
* Low professional status (blue collars)
* Being between 35-70 years
* Eligible to follow the given tasks

Exclusion Criteria:

* No volunteering to join to the study
* No eagerness to give information about his/her physical activity level
* Do not let to perform the physical assessments

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-05-25 (Estimated); Study Completion 2022-10-25 (Estimated)

PRIMARY OUTCOMES:
Physical measures | 4 months
  To understand the weight status of the participants will be assessed as weight in kilograms and height in meters; body mass index (as weight and height combined in kg/m2); and Ponderal Index (as weight and height combined in kg/cm) to understand if they are underweight, normal, heavy weight, obese, morbid obese; The waist circumference in centimetre to observe if it is above 95 cm for men and 80 cm for women is considered as higher than normal; if higher than 110cm for men and 88cm for women is considered as having risks for obesity, metabolic syndrome, diabetes, cardiovascular diseases.

SECONDARY OUTCOMES:
Hand and pinch grip power | 4 months
  Hand and pinch grip power will be assessed by an electronic dynamometer in Newton.
  If the elbow is in extension during hand grip this will provide the data on the power of upper extremity, and if it is flexed at 90 degrees and forearm is supported on the table, this provides handgrip power.
  The data will be compared with the normative data according to gender and the age groups of the participants.
Level of physical activity | 4 months
  The level of physical activity will be assessed by the International Physical Activity Questionnaire- IPAQ searching the amount of walking and low, moderate and high intensity physical activities as total time in minutes in days and frequency in days of week; Both activity and sitting behaviors will be measured if they perform at least once and not less than 10 minutes over the past 7 days.
  The scores will be achieved by the multiplication of the minutes, days and MET values in a week, as MET minutes/weeks.
  Walking score will be achieved by the multiplication of 3.3 METs with the total walking duration in minutes in a week; the total weekly walking duration will be multiplied with 4 METs for the medium level of walking and 8 METs for the vigorous level of walking.

CONTACTS AND LOCATIONS:
Overall Officials: Serap Inal, PhD, Principal Investigator — Istinye University
Locations (1):
- Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Uffelen JG, Wong J, Chau JY, van der Ploeg HP, Riphagen I, Gilson ND, Burton NW, Healy GN, Thorp AA, Clark BK, Gardiner PA, Dunstan DW, Bauman A, Owen N, Brown WJ. Occupational sitting and health risks: a systematic review. Am J Prev Med. 2010 Oct;39(4):379-88. doi: 10.1016/j.amepre.2010.05.024. PMID 20837291
- [Background] Tremmel M, Gerdtham UG, Nilsson PM, Saha S. Economic Burden of Obesity: A Systematic Literature Review. Int J Environ Res Public Health. 2017 Apr 19;14(4):435. doi: 10.3390/ijerph14040435. PMID 28422077
- [Background] Dunstan DW, Howard B, Healy GN, Owen N. Too much sitting--a health hazard. Diabetes Res Clin Pract. 2012 Sep;97(3):368-76. doi: 10.1016/j.diabres.2012.05.020. Epub 2012 Jun 9. PMID 22682948
- [Background] Neuhaus M, Healy GN, Dunstan DW, Owen N, Eakin EG. Workplace sitting and height-adjustable workstations: a randomized controlled trial. Am J Prev Med. 2014 Jan;46(1):30-40. doi: 10.1016/j.amepre.2013.09.009. PMID 24355669
- [Background] Shrestha N, Pedisic Z, Neil-Sztramko S, Kukkonen-Harjula KT, Hermans V. The Impact of Obesity in the Workplace: a Review of Contributing Factors, Consequences and Potential Solutions. Curr Obes Rep. 2016 Sep;5(3):344-60. doi: 10.1007/s13679-016-0227-6. PMID 27447869
- [Background] Judice PB, Hamilton MT, Sardinha LB, Zderic TW, Silva AM. What is the metabolic and energy cost of sitting, standing and sit/stand transitions? Eur J Appl Physiol. 2016 Feb;116(2):263-73. doi: 10.1007/s00421-015-3279-5. PMID 26467968